CLINICAL TRIAL: NCT03312257
Title: Myopia Control in Children With Low-dose Atropine and Soft Bifocal Contact Lenses
Brief Title: Bifocal & Atropine in Myopia (BAM) Study
Acronym: BAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenny Jones (Other)
Responsible Party: Sponsor-Investigator, Jenny Jones, Research Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23EY025273 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Atropine

ARMS (1):
- Multifocal D +2.50 add & 0.01% atropine (Experimental): The Biofinity Multifocal "D" with a +2.50 add is a soft bifocal contact lens that has a strong reading power; the 0.01% atropine is a low-dose atropine.
  Interventions: Combination Product: Multifocal D +2.50 add & 0.01% atropine

INTERVENTIONS:
Combination Product: Multifocal D +2.50 add & 0.01% atropine — Biofinity Multifocal D +2.50 add is a monthly disposable contact lens commercially available from CooperVision; 0.01% atropine is low-dose atropine compounded by local pharmacy.

SUMMARY:
This study will test whether the combined treatment of 0.01% atropine and soft bifocal contact lens wear produces slower myopia progression and axial elongation compared to soft bifocal contact lenses alone in children ages 7 to 11 years old.

DETAILED DESCRIPTION:
Both atropine and soft bifocal contact lenses have been shown to slow myopia progression, and both can cause changes in choroidal thickness. But the relationship between these mechanisms is unclear. The central hypothesis to be tested in the BAM Study is that atropine and soft bifocal contact lenses each exert their anti-progression actions through a common pathway that involves the choroid. If this is correct, then adding atropine treatment to soft bifocal contact lens wear will lead to a more effective slowing of myopia progression than prescribing soft bifocal contact lenses alone due to the additive effects in the common pathway.

The BAM Study is an ancillary study of an NIH sponsored multi-center, randomized clinical trial, the Bifocal Lenses In Nearsighted Kids (BLINK) Study (NIH: U10EY023208; NCT: NCT02255474). The BLINK Study compares myopia progression between subjects who wear single vision contact lenses and those wearing soft bifocal contact lenses. The BAM Study enrolls an additional 49 subjects that are age-matched with the participants who are wearing +2.50D add soft bifocal contact lenses in the BLINK Study. The subjects in the BAM Study wear +2.50D add soft bifocal contact lenses in combination with daily administration of one drop of 0.01% atropine in each eye for three years. The rates of myopia progression and axial elongation will be compared to the rates in participants who are receiving treatment with +2.50D add soft bifocal contact lenses alone in the BLINK Study.

Two specific aims will be addressed: Aim 1: To test whether the combined treatment of 0.01% atropine and soft bifocal contact lens wear produces slower myopia progression and axial elongation compared to soft bifocal contact lenses alone over 3 years. Aim 2: To test whether early changes in choroidal thickness can be used as predictors of long-term myopia progression / axial elongation. The results of this study will have significant implications for future studies to develop and test new therapeutic regimes that optimize the effect of myopia control through combined pharmacological and optical interventions. The outcomes will also aid in understanding the potential role of short-term changes of choroidal thickness in long- term regulation of myopia progression and ocular growth.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 11 years, inclusive, at baseline examination
* -0.75 to -5.00 D, inclusive, spherical component, cycloplegic autorefraction
* ≤1.00 DC, cycloplegic autorefraction
* ≤ 2.00 D difference between the sphere components of the two eyes (anisometropia), cycloplegic autorefraction
* 0.1 logMAR or better best-corrected visual acuity in each eye
* 0.1 logMAR or better visual acuity OU distance and near with a +2.50 D add contact lens
* +2.50 D add lens provides adequate fit with respect to movement and centration
* Finish at least 71% of 0.01% atropine during the run-in period

Exclusion Criteria:

* Eye disease or binocular vision problems (e.g., strabismus, amblyopia, oculomotor nerve palsies, corneal disease, etc.)
* Previous intraocular or corneal surgery
* Systemic disease that may affect vision, vision development, or contact lens wear (eg, diabetes, Down syndrome, etc.)
* Previous gas permeable, soft bifocal, or orthokeratology contact lens wear or bifocal/PAL spectacle wear (longer than 1 month of wear)
* Previous or current participation in myopia control studies
* Chronic use of medications that may affect immunity, such as oral or ophthalmic corticosteroids for ocular or systemic diseases
* Issues that may interfere with the ability to participate over the next 3 years

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Huang, PhD, OD, Principal Investigator — The Ohio State Univeristy

REFERENCES:
- [Derived] Jones JH, Mutti DO, Jones-Jordan LA, Walline JJ. Effect of Combining 0.01% Atropine with Soft Multifocal Contact Lenses on Myopia Progression in Children. Optom Vis Sci. 2022 May 1;99(5):434-442. doi: 10.1097/OPX.0000000000001884. Epub 2022 Feb 25. PMID 35511120
- [Derived] Huang J, Mutti DO, Jones-Jordan LA, Walline JJ. Bifocal & Atropine in Myopia Study: Baseline Data and Methods. Optom Vis Sci. 2019 May;96(5):335-344. doi: 10.1097/OPX.0000000000001378. PMID 31046016

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multifocal D +2.50 Add & 0.01% Atropine
Started | 49
Completed | 46
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Multifocal D +2.50 Add & 0.01% Atropine
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Refractive Error Progression
Description: Refractive error, as measured by cycloplegic autorefraction in both eyes, will be measured yearly to assess the difference in progression between the combination treatment (+2.50 D add soft bifocal lens and 0.01% atropine) group and the historical control group (+2.50 D add soft bifocal lens only) in the BLINK Study.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Multifocal D +2.50 Add & 0.01% Atropine
Number analyzed (Participants) | 46
Diopter | -3.50 (0.72)
Statistical Analysis 1: Comparison: Multifocal D +2.50 Add & 0.01% Atropine; Test type: Other — Repeated measures analyses using mixed linear models in STATA (version 15) were undertaken to model myopia progression (primary outcome) and axial elongation (secondary outcome) to account for the clusters of correlated data due to repeated participant outcome measures; p = 0.70, Repeated measures analyses; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.14 to 0.21]

2. Secondary Outcome: Axial Length Progression
Description: Axial length progression, as measured by Lenstar in both eyes, will be measured yearly to assess the difference in progression between the combination treatment (+2.50 D add soft bifocal lens and 0.01% atropine) group and the historical control group (+2.50 D add soft bifocal lens only) in the BLINK Study.
Time Frame: 3 years
Measure: Mean (Standard Error); unit: mm
Arm/Group | Multifocal D +2.50 Add & 0.01% Atropine
Number analyzed (Participants) | 46
mm | 22 (0.75)
Statistical Analysis 1: Comparison: Multifocal D +2.50 Add & 0.01% Atropine; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.054, Repeated measures analyses; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.16 to 0.002]

ADVERSE EVENTS:
Time Frame: Three years
Arm/Group | Multifocal D +2.50 Add & 0.01% Atropine
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 46/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Multifocal D +2.50 Add & 0.01% Atropine (N=46)
Mild eye itching at the drops administering site, which resolved within a few minutes per subjects. (Eye disorders) | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT03312257/Prot_SAP_000.pdf